CLINICAL TRIAL: NCT02445196
Title: PTSD Coach App Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Barr Taylor (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Craig Barr Taylor, Professor Emeritus, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22977
Record Dates: First submitted 2015-05-11; First posted 2015-05-15 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2016-12

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTSD Coach (Experimental): Subjects assigned to this condition receive information about how to download the research app, PTSD Explorer. This research version of PTSD Coach functions exactly the same, however we have the ability to track individual usage of the app. The app contains contains psycho-education about PTSD and the management of symptoms of PTSD along with activities and techniques to address symptoms. Subjects are told to use the app as much or as little as they want over the next three months.
  Interventions: Behavioral: PTSD Coach; Device: Smartphone
- Waitlist Control (Active Comparator): Subjects assigned to this condition are told: "You have been randomly assigned to Group 2, the group that does not use the app."
  Following their completion of the post-intervention assessment at 3 months, they are told how to access to the publicly available PTSD Coach app in the Apple App Store or Android Play Store, just so that they are made aware of the resources available to them.
  Interventions: Behavioral: PTSD Coach; Device: Smartphone

INTERVENTIONS:
Behavioral: PTSD Coach — PTSD Coach is a mobile app that aims to teach individuals self-management strategies for symptoms of PTSD.
Device: Smartphone — All participants must have a smartphone, either apple or android.

SUMMARY:
PTSD Coach is a mobile application (app) that aims to teach individuals self-management strategies for symptoms of Post-traumatic Stress Disorder (PTSD). PTSD is a major public health concern. Although effective treatments exist, affected individuals face many barriers to receiving traditional care. As smartphones are now carried by more than half of the U.S. population, they have the potential to overcome many of these barriers by delivering self-help interventions on apps. Despite PTSD Coach's use of evidence-based cognitive behavioral strategies there is still a need to test the effectiveness of the app in managing PTSD symptoms. This controlled, two-arm, randomized (1:1) trial will evaluate the efficacy, feasibility and acceptability of PTSD Coach to reduce PTSD symptoms in a community sample of trauma survivors with PTSD symptoms. After completing an eligibility phone screen or online screen, individuals who score a 35 or above on the PTSD Checklist (PCL) and consent will complete a baseline assessment and then be randomized to the PTSD Coach app condition or a waitlist control group. Additionally, those assigned to the PTSD Coach intervention will be instructed to download a research version of the app, called PTSD Explorer, that enables passive and objective monitoring of app use. Each individual will be reassessed at post-intervention (3 months) and follow-up (3 months later, or 6 months after completing baseline). The investigators predict that those using the PTSD Coach app will demonstrate a significant and sustained reduction in PTSD symptoms and increase in patient coping self-efficacy compared to the waitlist control group. The investigators will explore if there is a relationship between levels of engagement and PTSD symptom change.

ELIGIBILITY:
Inclusion Criteria:

1. Experienced or witnessed an extremely traumatic event that involved actual or threatened death or serious injury to you or someone else. Event must have occurred more than 1 month ago.
2. Significant PTSD symptoms. Total PTSD Checklist Score ≥ 35.
3. Have a smartphone or smart device that can download apps (iPhone, iPod touch, iPad, or android phone or tablet).
4. English is the primary language.
5. Available for the next 6 months to participate in the study and use smart device.

Exclusion Criteria:

1. Unable to give informed consent.
2. Is currently receiving mental health treatment.
3. Currently participating in other PTSD-related research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C Barr Taylor, M.D., Principal Investigator — Stanford University

RESULTS

PARTICIPANT FLOW:
Groups:
- Waitlist Control: Subjects assigned to this condition are told: "You have been randomly assigned to Group 2, the group that does not use the app."
  Following their completion of the post-intervention assessment at 3 months, they are told how to access to the publicly available PTSD Coach app in the Apple App Store or Android Play Store, just so that they are made aware of the resources available to them.
  PTSD Coach: PTSD Coach is a mobile app that aims to teach individuals self-management strategies for symptoms of PTSD.
  Smartphone: All participants must have a smartphone, either apple or android.
Period: Overall Study
Arm/Group | PTSD Coach | Waitlist Control
Started | 62 | 58
Completed | 51 | 52
Not Completed | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTSD Coach | Waitlist Control | Total
Number analyzed (Participants) | 62 | 58 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 57 | 115
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.43 (15.16) | 39.12 (14.08) | 39.28 (14.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 37 | 83
  Male | 16 | 21 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 58 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptoms Measured by the Post Traumatic Stress Disorder Checklist (PCL)
Description: PTSD symptoms were assessed with the PCL-C (Weathers et al., 1993), a 17-item self-report measure of DSM-IV PTSD symptoms with strong psychometric properties (Wilkins, Lang, & Norman, 2011). Items are rated on how much the symptom bothered the respondent in the past month on a scale ranging from 1 (not at all) to 5 (extremely), with the sum score ranging from 17 to 85 providing a symptom severity rating, with higher ratings indicating more severe PTSD symptoms.
Time Frame: Baseline to Posttreatment (3 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTSD Coach | Waitlist Control
Number analyzed (Participants) | 62 | 58
units on a scale
  Baseline | 63.19 (11.78) | 60.59 (10.24)
  Posttreatment | 51.93 (14.04) | 53.90 (13.78)
Statistical Analysis 1: Comparison: PTSD Coach vs Waitlist Control; Repeated measures ANOVAs assessed the condition by time (baseline to posttreatment) interaction effects covarying PTSD treatment. Following the ITT principle, data from all randomized participants were analyzed and multiple imputation replaced missing values. A power analysis indicated that to achieve 80% power to detect an effect size in the magnitude (i.e., d = 0.25 to .33) with alpha of .05 and a correlation between repeated measures of .5, 60 participants per condition would be needed; Test type: Superiority or Other; p = .035, ANOVA; Mean Difference (Net) = 4.57

2. Secondary Outcome: Change in Subject Coping Self-efficacy Measured by a Questionnaire Assessing Confidence in Managing Core Symptoms of PTSD Addressed in the Intervention
Description: PTSD symptom coping SE was assessed with a 9-item self-report measure developed for the study following Bandura's guidelines (Bandura, 2006). Items assess confidence in managing PTSD symptoms and reaching out for support on a scale from 0 (cannot do at all) to 100 (highly certain can do). The average score provides an overall measure of SE with higher scores reflecting greater self-efficacy coping with PTSD symptoms. Cronbach's alpha at baseline was .87.
Time Frame: Baseline to Posttreatment (3 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTSD Coach | Waitlist Control
Number analyzed (Participants) | 62 | 58
units on a scale
  Baseline | 49.63 (19.28) | 50.77 (19.10)
  Posttreatment | 56.09 (18.35) | 52.36 (19.16)
Statistical Analysis 1: Comparison: PTSD Coach vs Waitlist Control; Test type: Superiority or Other; p = .086, ANOVA; Mean Difference (Net) = 4.87

3. Secondary Outcome: Change in Interpersonal Functioning Measured by a Brief Inventory of Psychosocial Functioning (IPF7)
Description: Psychosocial functioning was measured using the Brief Inventory of Psychosocial Functioning (B-IPF; Erb, Kearns, Bovin et al., 2015), a 7-item self-report measure. Items are rated on how much trouble the respondent had in the past month in relationships or other important areas of functioning (e.g., work, training or education) on a scale ranging from 0 (not at all) to 6 (very much). An average of applicable items provides an index of psychosocial functioning, with higher scores reflecting more poorer psychosocial functioning. Cronbach's alpha at baseline was .82.
Time Frame: Baseline to Posttreatment (3 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTSD Coach | Waitlist Control
Number analyzed (Participants) | 62 | 58
units on a scale
  Baseline | 3.85 (1.55) | 3.15 (1.40)
  Posttreatment | 2.86 (1.47) | 2.91 (1.49)
Statistical Analysis 1: Comparison: PTSD Coach vs Waitlist Control; Test type: Superiority or Other; p = .007, ANOVA; Mean Difference (Net) = 0.75

4. Secondary Outcome: Change in Depression Symptoms Measured by the Patient Health Questionnaire (PHQ8)
Description: Depression was assessed with the Patient Health Questionnaire depression scale (PHQ-8; Kroenke et al., 2009), an 8-item self-report measure of depression with evidence showing its ability to measure depression symptom severity and potential diagnosis. Items are rated on how much the symptom bothered the respondent in the past two weeks on a scale ranging from 0 (not at all) to 3 (nearly every day). Total scores can range from 0 to 24, with higher scores indicating more severe depression symptoms. Cronbach's alpha at baseline was .87.
Time Frame: Baseline to Posttreatment (3 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTSD Coach | Waitlist Control
Number analyzed (Participants) | 62 | 58
units on a scale
  Baseline | 15.06 (6.36) | 13.62 (5.55)
  Posttreatment | 11.03 (5.29) | 12.31 (5.88)
Statistical Analysis 1: Comparison: PTSD Coach vs Waitlist Control; Test type: Superiority or Other; p = .005, ANOVA; Mean Difference (Net) = 2.72

5. Secondary Outcome: Sustained Change in PTSD Symptoms Measured by the Post Traumatic Stress Disorder Checklist (PCL)
Description: as for outcome 1
Time Frame: Postreatment to 3-month Follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTSD Coach
Number analyzed (Participants) | 62
units on a scale
  Posttreatment | 51.93 (14.04)
  3-Month Follow-up | 49.15 (13.94)
Statistical Analysis 1: Comparison: PTSD Coach; Test type: Superiority or Other; p = .113, t-test, 2 sided; Mean Difference (Net) = 2.78

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | PTSD Coach | Waitlist Control
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/58
Other Adverse Events (participants affected / at risk) | 0/62 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No